CLINICAL TRIAL: NCT04664374
Title: Characterizing MyMood Patterns of Use
Status: Active, not recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. David Kreindler, Head, Division of Youth Psychiatry, Sunnybrook Health Sciences Centre
Other Study IDs: 396-2019
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Bipolar Disorder; Mood Disorders; Depression; Dysthymia
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Depression; Dysthymic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mood Disorder: Based on screening questions administered on-line as part of the enrollment process, participants will be divided into two groups: (i) those who screen positive for a history of mood disorders and (ii) all other participants. All outcome measures apply only to the mood disorder group.
  Interventions: Other: MyMood
- Other: see above
  Interventions: Other: MyMood

INTERVENTIONS:
Other: MyMood — Users will use the MyMood tool. Each MyMood session consists of a brief survey, followed by a few psycho-educational 'tips'(targeted psycho-educational interventions received from time to time based on symptom severity reports as determined by the software algorithm).

SUMMARY:
MyMood is an electronic mood-charting tool available to the general population of Sunnybrook Health Sciences Centre (SHSC). This project aims to characterize duration and frequency of use of MyMood by users characteristics and determine if there is any significant variability in duration and frequency of use attributable to users' age, sex, self-reported diagnosis of a mood disorder, and/or prior treatment.

DETAILED DESCRIPTION:
Mental Health Telemetry (MHT) is a software platform developed at Sunnybrook for collecting real-time self-report symptom-rating questionnaire data using patients' cell phones or other portable, Internet-enabled devices. MHT has previously been used in several funded clinical research studies. The mood-disorders-specific version of MHT, which we have named MyMood, collects information on a variety of items including symptom severity, medication adherence, ER visits / hospital admissions, sleep, relationships, and life events. In our previous project, we made MyMood available to the general population of SHSC by integrating it into Sunnybrook's MyChart personal health record system and collected feedback from users, using the feedback to refine MyMood. In the current project, we aim to characterize long-term patterns of MyMood usage, examining how duration and frequency of use are affected by demographic and clinical characteristics of users (age, sex, present / reported diagnosis of a mood disorder, and/or prior treatment).

Please note that the _only_ route for entry into this study is self-referral: interested individuals who have signed themselves up for MyChart can choose to begin using MyMood on their own. There is no reason to contact the study team regarding recruitment.

ELIGIBILITY:
Inclusion Criteria:

• Registered user of Sunnybrook Health Sciences Centre "MyChart" electronic patient portal

Exclusion Criteria:

• n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Registered user of Sunnybrook Health Sciences Centre "MyChart" electronic patient portal
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2025-01-06 (Estimated); Study Completion 2025-01-06 (Estimated)

PRIMARY OUTCOMES:
MyMood Use | 3 years
  Number of MyMood reports generated per user per month

CONTACTS AND LOCATIONS:
Overall Officials: David M Kreindler, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada